CLINICAL TRIAL: NCT02416466
Title: Phase Ib Trial of CAR-T Hepatic Artery Infusions Followed by Selective Internal Radiation Therapy (SIRT) With Yttrium-90 Sir-Spheres® for CEA-Expressing Liver Metastases
Brief Title: CAR-T Hepatic Artery Infusions and Sir-Spheres for Liver Metastases
Acronym: HITM-SIR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roger Williams Medical Center (Other)
Collaborators: Sirtex Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 383-74
Record Dates: First submitted 2015-03-30; First posted 2015-04-15 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Liver Metastases
Keywords: Colorectal cancer; Liver metastases; Breast cancer; Gastric cancer; Pancreas cancer; Carcinoembryonic antigen; CAR-T; Immunotherapy
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- anti-CEA CAR-T cells + Sir-Spheres (Experimental): Three infusions of gene-modified anti-CEA T cells over the course of 6 weeks into the hepatic artery via a percutaneous approach along with low dose IL-2. A single dose of Sir-Spheres will be given 2 weeks following the final T cell dose.
  Interventions: Biological: anti-CEA CAR-T cells; Device: Sir-Spheres

INTERVENTIONS:
Biological: anti-CEA CAR-T cells — Gene modified patient T cells.
  Other Names: Designer T cells
Device: Sir-Spheres — SIR-Spheres microspheres are a medical device used in Selective Internal Radiation Therapy (SIRT) for liver tumors. SIR-Spheres microspheres are a permanent implant and for single use only. The biocompatible resin microspheres containing yttrium-90 have a median diameter of 32.5 microns (range between 20 and 60 microns).
  Other Names: Selective Internal Radiation Therapy (SIRT); Yttrium-90 microspheres

SUMMARY:
This is an open label fixed dose phase Ib of anti-CEA CAR-T cells hepatic artery infusions and yttrium-90 SIR-Spheres in patients with CEA-expressing liver metastases.

DETAILED DESCRIPTION:
Patients undergo leukapheresis from which peripheral blood mononuclear cells are purified. T cells are activated and then re-engineered to express chimeric antigen receptors (CARs) specific for CEA. Cells are expanded in culture and returned to the patient by percutaneous hepatic artery infusion at specific cell doses. Prior to the first dose, each patient will undergo diagnostic angiography to verify suitable arterial anatomy. Three anti-CEA CAR-T doses and one SIR-Sphere dose per patient are planned at 2-week intervals. Low dose interleukin-2 will be given via an ambulatory infusion pump for 6 weeks.Normal liver and tumor biopsies will be obtained at the time of the initial diagnostic angiogram and during the final infusion session.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically confirmed diagnosis of CEA+ adenocarcinoma and liver metastases. Patient must have either histologic confirmation of the liver metastases or histologic documentation of the primary tumor and definitive radiologic evidence of liver involvement. Measurable disease is required with lesions of > 1.0 cm by CT. Soluble CEA is not acceptable as the sole measure of disease. Limited extrahepatic disease is acceptable if confined to the lungs or peritoneal cavity.
* Tumor must be CEA-expressing as demonstrated by elevated serum CEA levels (≥10ng/ml) or immunohistochemistry on a biopsy specimen. Archived tissue is acceptable for determination of CEA expression.
* Patient must be at least 18 years of age.
* Patient able to understand and sign informed consent.
* Patient with a life expectancy of greater than four months.
* Patient failed at least one line of standard systemic chemotherapy and has unresectable disease.
* Patient with performance status of 0 to 1 (ECOG).
* Patient with adequate organ function as defined in protocol.
* Acceptable hepatic vascular anatomy as determined by CT, MR, or conventional angiography. A nuclear medicine study will be performed to document the absence of a significant hepatic-pulmonary shunt (<20%).

Exclusion Criteria:

* Female patients of childbearing age will be tested for pregnancy. Pregnant patients will be excluded from the study. Males who are actively seeking to have children will be made aware of the unknown risks of this study protocol on human sperm and the need to practice birth control.
* Patients with serious or unstable renal, hepatic, pulmonary, cardiovascular, endocrine, rheumatologic, or allergic disease based on history, physical exam and laboratory tests will be excluded, as outlined in section 5.2.8.
* Patients with active clinical disease caused by CMV, hepatitis B or C, HIV or tuberculosis will be excluded from the study.
* Patients who have had cytotoxic and/or radiation therapy within 4 weeks prior to entry into the trial or 4 weeks prior to infusion will be excluded. Patients with other concurrent malignancies will be excluded.
* Patients requiring systemic steroids will be excluded.
* Patients with unsuitable hepatic vascular anatomy will be excluded from the study.
* Patients with extrahepatic metastatic disease beyond the lungs or abdominal/ retroperitoneal lymph nodes.
* Patients with >50% liver replacement at time of treatment will be excluded.
* Previous external beam radiotherapy to the liver.
* Portal vein thrombosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-04; Primary Completion 2016-11-21 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Safety of CAR-T cell hepatic artery infusions in combination with Sir-Spheres as Measured by Number of Participants with Adverse Events | 14 weeks
  To determine the safety and regimen limiting toxicity (RLT) of a standard of care treatment with Yttrium-90 Sir-Spheres Microspheres when following anti-CEA CAR-T hepatic artery infusions (HAI) for CEA-expressing liver metastases.

SECONDARY OUTCOMES:
Treatment response (Liver tumor response by MRI, PET, CEA level, and biopsy) | 14 weeks
  Liver tumor response by MRI, PET, CEA level, and biopsy
  1. RECIST and immune related response criteria (MRI & PET)
  2. By evidence of tumor necrosis and fibrosis (biopsy)
Serum cytokine levels | 14 weeks
  Measurement of cytokines as indicators of immune response
CAR-T detection in liver tumors, normal liver, and extrahepatic sites | 14 weeks
  Quantification of CAR-T cells in biopsy and blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Steven C Katz, MD, Principal Investigator — Roger Williams Medical Center
Locations (1):
- Roger Williams Medical Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No